CLINICAL TRIAL: NCT03224702
Title: A Single-Center, Phase I, Randomized, Double Blind, Placebo-Controlled, First-In-Human Trial to Assess the Safety, Tolerability, Immunogenicity, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of Subcutaneous Injected M6495 (Anti-ADAMTS-5 Nanobody) in Healthy Male Subjects
Brief Title: First-in-Human Trial of Anti-ADAMTS-5 Nanobody in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS200572-0009; 2017-001663-21 (EudraCT Number)
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Healthy
Keywords: M6495; anti-A disintegrin and metalloproteinase with thrombospondin motifs-5 nanobody; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M6495 (Experimental)
  Interventions: Drug: M6495
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: M6495 — Subjects will receive M6495 on Day 1
  Arms: M6495
Drug: Placebo — Subjects will receive placebo matched to M6495 on Day 1
  Arms: Placebo

SUMMARY:
This First-In-Human trial will be conducted in healthy male subjects to explore the safety, tolerability, immunogenicity, pharmacokinetics, and pharmacodynamics of single doses of M6495.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Body Mass Index (BMI) of greater than or equal to (>=) 18.5 and less than or equal to (=<) 29.9 Kilogram per square meter (kg/m^2), and a body weight between 50 and 100 kg at screening.
* Subjects must agree to use effective method(s) of contraception during the trial.
* Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

* Subjects who have recently participated in other clinical trials.
* Donated blood, have a significant medical condition, history of drug hypersensitivity, consumption of large amounts of xanthine-containing foods or beverages, recent or ongoing concomitant medication, hypertension, tachycardia and significant findings on electrocardiogram
* Positive drug screening test, positive test for Hepatitis B or C or human immune deficiency virus (HIV), or have been kept in detention
* Other protocol defined exclusion criteria could apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-08-06 (Actual); Study Completion 2018-08-06 (Actual)

PRIMARY OUTCOMES:
Occurrence of Treatment-emergent Adverse Events (TEAEs) and Serious AEs (SAEs) | Baseline up to Day 75
Occurrence of TEAEs and SAEs by Severity | Baseline up to Day 75
Number of Subjects With Injection Site Reactions (ISRs) | Baseline up to Day 75
Number of Subjects with Clinically Significant Change From Baseline in Vital Signs, Laboratory Parameters and 12-lead Electrocardiogram (ECG) Findings | Baseline up to Day 75

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of M6495 | Pre-dose and 6, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, 168, 240, 336, 504, 672, 912, 1152, 1440, 1776 hours post-dose
Time to Reach Maximum Observed Serum Concentration (Tmax) of M6495 | Pre-dose and 6, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, 168, 240, 336, 504, 672, 912, 1152, 1440, 1776 hours post-dose
Area Under the Concentration-Time Curve From Time Zero to the Last Sampling Time (t) at Which the Concentration is at or Above the Lower Limit of Quantification (AUC0-t) of M6495 | Pre-dose and 6, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, 168, 240, 336, 504, 672, 912, 1152, 1440, 1776 hours post-dose
Area Under the Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of M6495 | Pre-dose and 6, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, 168, 240, 336, 504, 672, 912, 1152, 1440, 1776 hours post-dose
Apparent Terminal Half-Life (t1/2) of M6495 | Pre-dose and 6, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, 168, 240, 336, 504, 672, 912, 1152, 1440, 1776 hours post-dose
Apparent Terminal Rate Constant (λz) of M6495 | Pre-dose and 6, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, 168, 240, 336, 504, 672, 912, 1152, 1440, 1776 hours post-dose
Apparent Body Clearance (CL/F) of M6495 | Pre-dose and 6, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, 168, 240, 336, 504, 672, 912, 1152, 1440, 1776 hours post-dose
Apparent Volume of Distribution During the Terminal Phase (Vz/F) of M6495 | Pre-dose and 6, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, 168, 240, 336, 504, 672, 912, 1152, 1440, 1776 hours post-dose
Percent Change From Baseline in Serum Aggrecan Degradation neo-Epitope (ARGS) at Day 1, 2, 3, 4, 5, 6, 7, 8, 11, 15, 22, 29, 39, 49, 61 and 75 | Baseline, Day 1, 2, 3, 4, 5, 6, 7, 8, 11, 15, 22, 29, 39, 49, 61 and 75
Number of Subjects With Anti-drug Antibodies (ADA) for M6495 | Pre-dose, Day 8, 22, 49 and 75
Levels of Anti-Drug Antibodies (ADA) Titers | Pre-dose, Day 8, 22, 49 and 75
Change From Baseline in Telemetry Electrocardiogram (ECG) Intervals Up to 24 hours post Day 1 dose | Baseline, Up to 24 hours post Day 1 dose
Slope of Exposure vs QTc From Digital Electrocardiogram Triplicates | Baseline up to Day 75
Maximal Effect (Imax) of M6495 | Pre-dose and 6, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, 168, 240, 336, 504, 672, 912, 1152, 1440, 1776 hours post-dose
Inhibitory Concentration (IC) 10, IC50 and IC90 of M6495 | Pre-dose and 6, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, 168, 240, 336, 504, 672, 912, 1152, 1440, 1776 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- DanTrials ApS c/o Bispebjerg Hospital, Copenhagen, Denmark